CLINICAL TRIAL: NCT05353881
Title: Striatal Dopamine Transmission and Prodromal Markers of α-synucleinopathy Neurodegeneration in Recurrent Dream Enactment Behaviors Without REM Sleep Without Atonia: a Case-control Study
Brief Title: Prodromal Markers in Recurrent Dream Enactment Behaviors Without REM Sleep Without Atonia
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: RGC14107520
Record Dates: First submitted 2021-12-21; First posted 2022-04-29 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: REM Sleep Behavior Disorder
Keywords: Striatal dopamine; REM sleep without atonia; Prodromal markers
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
REM sleep behavior disorder is a novel and distinct parasomnia characterized by recurrent dream enactment behaviors (DEBs) and REM sleep without atonia (RSWA) during polysomnographic assessment, with a male predominance and typical onset age at early 60's. The majority of patients with idiopathic RBD (iRBD) will eventually develop α-synucleinopathy, for instance Parkinson's disease (PD). Thus, iRBD has been considered as a highly specific precursor of α-synucleinopathy-related neurodegeneration. Recently, increasing studies have found that some participants present with only RSWA or DEBs (but without sufficient RSWA), which does not meet the diagnostic criteria for RBD. It has been suggested that these participants with subclinical features (either DEBs or RSWA) might represent a condition known as prodromal RBD. Several emerging evidence, including our own study, have implied a link between isolated RSWA (RSWA without DEBs) and markers of α-synucleinopathy-related neurodegeneration. However, it is still unclear whether the other condition related to RBD, i.e. recurrent DEBs but without sufficient RSWA, is related to a certain degree of α-synucleinopathy. In this regard, the novel concept of recurrent DEBs but without sufficient RSWA, also termed as prodromal/isolated RBD by some researchers, requires validation by further evidence in terms of clinical feature and neurodegenerative prodromal markers perspectives.

DETAILED DESCRIPTION:
This proposed study is a case-control study, which aims to determine whether recurrent DEBs but without sufficient RSWA represents an early stage of α-synucleinopathy. The investigators will recruit 62 participants with recurrent DEBs but without sufficient RSWA and their age-, sex- matched controls from the community and on-going projects. All participants will undergo clinical interview, comprehensive measures of prodromal markers of neurodegeneration (including excessive daytime sleepiness, olfactory functioning, constipation, erectile dysfunction, urinary dysfunction, symptomatic hypotension, depression, and clinical motor markers) as suggested by the International Parkinson and Movement Disorder Society (MDS) research criteria. In addition, a subset of the sample (n = 26 in each group) will undergo the triple-tracer positron emission tomography/computed tomography (PET/CT) imaging protocol of 18F-DOPA, to determine dopamine functions in putamen. This proposed study will help to disentangle the core features of RBD and validate the concept of prodromal RBD with reference to prodromal markers related to α-synucleinopathy neurodegeneration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 65 years old
* RBDQ-HK behavior factor greater > 8
* Recurrent DEBs by interview and/or video analysis
* Absence of sufficient RSWA

Exclusion Criteria:

* Age- and sex- matched with cases
* RBDQ-HK behavior factor < 8
* No DEBs by either interview or video analysis
* Absence of sufficient RSWA

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruiting ability for the current study is further evidenced by a series of studies and publications in the past few years. For example, in our ongoing case-control family study, the investigator have recruited 89 control proband and 64 their FDRs who have all underwent v-PSG (Liu et al, Annals of Neurology 2019). By now, the investigator have expanded the number to 103 control probands and 91 FDRs. The investigator believe that this cohort will help us to recruit sufficient number of control subjects in this proposed study.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Parkinson's Disease | 1 year
  overall probability of prodromal PD based on the MDS research criteria for prodromal PD

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kwok Wing, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Shatin Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
In this stage, we didn't decide which information of IPD will be share with other researchers